CLINICAL TRIAL: NCT06074055
Title: PREFER: PRogrammed Versus Modified Natural Cycle After Euploid Failed Embryo Transfer: A Randomized Control Trial
Brief Title: PRogrammed Versus Modified Natural Cycle After Euploid Failed Embryo Transfer
Acronym: PREFER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment issues
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2302-BRG-024-ES
Record Dates: First submitted 2023-09-20; First posted 2023-10-10 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Programmed FET Protocol (Other): Patients in this arm of the study will proceed with another programmed FET protocol which involves taking exogenous estrogen by mouth to stimulate the uterine lining to grow and develop. Once the lining has reached ≥ 7 mm and an endometrial pattern of type 1 or type 2, intramuscular progesterone in oil (50mg/ml daily) will be started at 8am on the morning that progesterone is initiated and continued per routine.
  Interventions: Other: FET Protocol
- Modified Natural FET Protocol (Other): Following development of at least one dominant follicle and endometrial proliferation ≥ 7 mm during cycle monitoring, patient will undergo administration of human chorionic gonadotropin (hCG) trigger shot followed by initiation of vaginal progesterone administration in accordance with institutional protocols.
  Interventions: Other: FET Protocol

INTERVENTIONS:
Other: FET Protocol — Participants are randomized to either another programmed FET Protocol vs. a modified natural FET protocol

SUMMARY:
The goal of this randomized clinical trial is to compare frozen embryo transfer protocols in patients undergoing a second frozen embryo transfer (FET) after a unsuccessful first programmed FET cycle as a possible treatment for people undergoing infertility treatment.

The purpose of this research study is to:

* Determine if there is a difference between FET protocols in patients who require a second FET cycle.
* Investigate if switching the FET protocol after a failed programmed cycle is beneficial for patients undergoing a second FET cycle.
* Examine pregnancy outcomes including obstetrical and neonatal outcomes (if applicable)
* Obtain uterine flexibility/stiffness measurements via transvaginal ultrasound prior to the embryo transfer procedure. This is called shear wave elastography.

Participants will be randomized in their second FET transfer attempt to either another programmed protocol or a modified natural protocol.

DETAILED DESCRIPTION:
This research study is studying if there is a difference in frozen embryo transfer protocols used (modified natural versus programmed) after a failed first programmed FET cycle, defined as either a negative pregnancy test or a biochemical loss, as a possible treatment for people undergoing infertility treatment and in vitro fertilization (IVF). Participants will be randomized, in a 1:1 ratio, in their second FET transfer attempt to either another programmed protocol or a modified natural protocol. Once randomized, participants will undergo routine FET monitoring based on their randomization allocation, transfer procedure and pregnancy monitoring as applicable. Additional ultrasound images will be obtained prior to the transfer procedure to assess the stiffness or flexibility of the uterus, called shear wave elastography. A participant blood sample and infant buccal swab will be collected for future research studies.

ELIGIBILITY:
Major Inclusion Criteria: The following are major inclusion criteria:

1. Patients planning to undergo frozen embryo transfer cycle with a single euploid blastocyst.
2. Patients who have previously undergone their first unsuccessful frozen embryo transfer cycle, defined as either failure of implantation with negative pregnancy test or biochemical pregnancy, using a programmed cycle protocol.
3. Preimplantation genetic testing for aneuploidy (PGT-A) of the embryo used in failed programmed embryo transfer cycle must have occurred after January 1, 2017.
4. Patients ages 18 to 53 years old as per practice guidelines.
5. Patients with BMI between 16-45 kg/m2.
6. Patients with at least one embryo remaining in storage, from either the same or a separate cohort.
7. Patients with proven ovulatory function, as defined by the presence of regular menstrual cycles or detection of luteinizing hormone surge on serum or urinary test kits.
8. Patients with ≥ 7 mm endometrial thickness prior to progesterone start in prior transfer cycle.
9. Normal uterine cavity as evidenced by recent (within 1 year) saline sonogram or hysteroscopy.

Major Exclusion Criteria: The following are exclusion criteria:

1. More than 1 prior unsuccessful frozen embryo transfer cycle.
2. The prior FET failure having had resulted in a clinical loss or ectopic pregnancy
3. Previously cancelled frozen embryo transfer cycle for inadequate endometrial response.
4. Patients who required a different route of estrogen administration in the prior programmed cycle (vaginal, transdermal, intramuscular).
5. PGT-A analysis of the available embryo for transfer performed prior to January 1, 2017.
6. Anovulatory or oligo-ovulatory patients unable to undergo modified natural endometrial preparation.
7. Patients with an endometrial thickness < 7 mm prior to progesterone start in prior cycle.
8. History of hypertensive disorders of pregnancy, including gestational hypertension, preeclampsia, and eclampsia.
9. Mullerian anomalies, excluding arcuate uterus and repaired septum.
10. No euploid embryos available for transfer.
11. Concurrent submucosal fibroids, unrepaired uterine defects or present indication for uterine surgery.
12. Communicating hydrosalpinx without plans for surgical correction prior to study enrollment.
13. Failure of patient to agree to enrollment in study with written consent.
14. Concurrent pregnancy.
15. Concomitant use of adjunctive therapies for endometrial proliferation or receptivity, including anticoagulation and antihistamines. These must be discontinued upon enrollment.
16. Embryo planned to be used for transfer generated from surgically obtained sperm.
17. Recurrent/persistent endometrial fluid in prior cycles visualized on the majority of transvaginal ultrasound monitoring.
18. Third party reproduction patients (donor sperm sources can be included).

Ages: 18 Years to 53 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Sustained implantation rate | approximately 6 weeks after embryo transfer
  presence of an intrauterine clinical pregnancy with fetal heart tones at 8 weeks gestational age

SECONDARY OUTCOMES:
Biochemical Pregnancy Rate | approximately 9 days after transfer
  Biochemical (positive serum beta human chorionic gonadotropin (bHCG) post transfer procedure)
Biochemical pregnancy loss rate | typically 1 month post initial bHCG test
  serum bHCG level ≥ 5 milli-International unit (mIU/mL) after FET without any ultrasound evidence of pregnancy until serum bHCG is < 5 mIU/mL
Clinical Pregnancy Rate | approximately 10 days after initial pregnancy test
  presence of an intrauterine gestational sac
Clinical Pregnancy Loss Rate | approximately 2 months after FET procedure
  a pregnancy after FET that had at minimum ultrasound evidence of a gestational sac, but did not progress to a live birth and was not terminated nor was an ectopic pregnancy.
Live Birth Rate | approximately 16-32 weeks post discharge at 8 weeks gestational age
  delivery of a live born infant greater than 24 weeks gestational age.
Rate of pregnancies of undetermined location and ectopic pregnancies | approximately 1-2 months post initial bHCG
  Pregnancies that are not intrauterine
Rate of maternal obstetrical outcomes and complications | approximately 40 weeks gestation
  mode of delivery, placental issues, preterm delivery
Rate of neonatal outcomes and complications | approximately 40 weeks gestational age or after delivery of infant
  gestational age at delivery, birth weight, any complications
Elastography Data | prior to the embryo transfer procedure
  shear wave elastography measurements of the uterus

CONTACTS AND LOCATIONS:
Overall Officials: Emre U Seli, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (2):
- United States (2):
  - Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey
  - Reproductive Medicine Associates of New Jersey, Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: No